CLINICAL TRIAL: NCT00706485
Title: Intra-Operative Dural Brachytherapy With Yttrium-90 Plaque Applicators
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New device for dural plaque irradiation was approved by FDA.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Implant Sciences (Unknown)
Responsible Party: Principal Investigator, Tom DeLaney, MD, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-007
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Spinal Neoplasms
Keywords: Y-90 plaque applicator; dural brachytherapy
MeSH Terms: conditions — Spinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dural brachytherapy plaque (Experimental): Patients undergoing spine tumor resection will undergo dural plaque brachytherapy.
  Interventions: Device: Yttrium-90 Plaque Applicator

INTERVENTIONS:
Device: Yttrium-90 Plaque Applicator — Placed on the dura during surgery for 10-17 1/2 minutes
  Other Names: Y-90 Plaque applicator

SUMMARY:
The purpose of this clinical trial is to determine the feasibility of the Y-90 plaque applicator. The Y-90 plaque application is designed to deliver high doses of radiation to tumors in the spine that involve dura (the tough outer layer of the spinal cord). Tumors in the spine need a high dose of radiation to kill cancer cells. The nearby spinal cord is a sensitive area which does not safely tolerate high doses of radiation. The Y-90 plaque applicator is a special technique used to deliver the radiation dose to the tumor cells and avoid the spinal cord.

DETAILED DESCRIPTION:
* The surgeon will remove the participants tumor from the outer layer of the spinal cord (dura). The Y-90 applicator and a "dummy" applicator will be brought to the surgery table in a protected container. A "dummy" applicator is the same size and shape as the Y-90 plaque applicator but does not contain radioactive plaque. The "dummy" applicator will be placed on the participants dura to make sure it fits properly, then it will be removed. The working Y-90 applicator will be placed on the dura for 10-17 1/2 minutes and then be removed.
* External beam irradiation is a type of high-energy radiation used to kill cancer cells and shrink tumors. This radiation will be given to the participant only if they have not had it prior to the study.
* After the treatment, participants will be asked to return for a follow-up visit 6 weeks, 3 months, every 6 months thereafter for 4 years, then annually to year 10. At these visits, they will have the following: physical examination; recent medical history; MRI or CT scan (twice each year) and; chest x-ray or chest CT (twice each year).

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of malignant tumor involving spine with extraosseous extension or arising in paraspinal soft tissues with tumor involving or abutting the dura. Patients with a limited metastatic disease and tumor involving the spine or paraspinal soft tissues and who are judged to benefit from surgery will also be eligible.
* Lesion may be primary or recurrent after prior surgery
* No clinical, radiographic or other evidence of distant metastatic tumor
* Fit for receiving the planned radiation dose to the affected site. No known genetic disease or medical condition associated with an abnormal radiation sensitivity.
* 18 years of age or older
* KPS of 70 or greater (excluding consideration of poor function due to the local growth or systemic metabolic effects of the tumor

Exclusion Criteria:

* Disease/conditions characterized by high radiation sensitivity
* Pregnancy
* Evidence of cord/cauda malfunction for causes other than effect os local tumor growth or due to metabolic effects of tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F. DeLaney, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dural Brachytherapy Plaque
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dural Brachytherapy Plaque
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Titanium-enclosed and Differentially-loaded Y-90 Dural Brachytherapy Plaque Fabrication and Use
Time Frame: At time of procedure
Measure: Number; unit: participants
Arm/Group | Dural Brachytherapy Plaque
Number analyzed (Participants) | 5
participants | 5

2. Secondary Outcome: Number of Participants With Local Control
Description: Local failure is defined as: extension of the tumor margin[s] in any direction at least 5 mm beyond that present on the pre-treatment imaging studies or the appearance of -tumor in tissues previously scored as sites of sub-clinical disease. Local control is absence of local failure.
Time Frame: at 6 weeks and at three months after therapy, and every 6 months thereafter for four years, and then annually to year 10
Measure: Number; unit: participants
Arm/Group | Dural Brachytherapy Plaque
Number analyzed (Participants) | 5
participants | 5

3. Secondary Outcome: Marginal Failure.
Description: Marginal failure is defined as appearance of tumor growth at the margin of dural plaque.
Time Frame: up to 10 years
Population: Study was closed without analysis of anatomic sites of failure. No data were collected for this outcome.
Arm/Group | Dural Brachytherapy Plaque
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Dural Brachytherapy Plaque
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes